CLINICAL TRIAL: NCT06173024
Title: Post Trial Access for Study SHP677-304: Recombinant Von Willebrand Factor (rVWF) for Adult and Pediatric Subjects With Severe Von Willebrand Disease (VWD)
Brief Title: Post Trial Access Program of TAK-577 for Von Willebrand Disease (VWD)
Status: Available | Type: Expanded Access
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-577 PTA
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Von Willebrand Disease (VWD)
Keywords: Drug Therapy
MeSH Terms: conditions — von Willebrand Diseases

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Biological: TAK-577 — TAK-577 as IV injection at dose calculated based on the participant's body weight.
  Other Names: Recombinant von Willebrand factor (rVWF); Vonvendi; Vonicog alfa; VEYVONDI

SUMMARY:
The post-trial access program allows eligible participants to gain access to unlicensed treatment on compassionate grounds. Recombinant von Willebrand factor (rVWF) also known as TAK-577, is a medicine to help treat Von Willebrand Disease (VWD). This post-trial access program enables continued access to children and adults who are benefitting from treatment on study SHP677-304 (NCT03879135) study.

DETAILED DESCRIPTION:
This is a post-trial access program in which the drug being given is called TAK-577. This study will provide access to TAK-577 before marketing authorization for eligible participants with severe VWD who are benefitting from treatment on study SHP677-304 and cannot adequately be treated via the current standard of care and cannot enter a clinical trial.

All participants will receive TAK-577 as a sequential intravenous infusion based on their weight.

This is a multi-center, international program. Participants will continue treatment until a benefit is no longer derived from the treatment (or treatment is no longer tolerable), the sponsor decision to end the program, the participant chooses to discontinue the treatment, or TAK-577 becomes commercially available for children.

ELIGIBILITY:
Inclusion Criteria:

1. Participant has completed the treatment period of the SHP677-304 study (at least 12 months on study treatment).
2. Participant had good clinical response to rVWF treatment.
3. Participant does not have access to any comparable or satisfactory alternative replacement therapy available at country level.
4. Participant will be/has been negatively impacted by discontinuation of rVWF.
5. Participant and/or a parent(s)/legal guardian is informed of the nature of the post-trial access program and can provide written informed consent for themselves or the child to participate (with assent from a child when appropriate) before treatment).

Exclusion Criteria:

1. Participants with known hypersensitivity/intolerance to the study drug will not be eligible for this study

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda

REFERENCES:
- See also: To obtain more information about this study, click this link — https://clinicaltrials.takeda.com/study-detail/19524029ced045e9?idFilter=%5B%22TAK-577+PTA%22%5D